CLINICAL TRIAL: NCT04622774
Title: A Phase 1/2, First-in-Human, Open-Label, Dose-Escalation and Expansion Study of IMGC936 (Anti-ADAM9 Antibody Drug Conjugate) in Patients With Advanced Solid Tumors
Brief Title: First-in-Human Study of IMGC936 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Collaborators: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMGC936-0901
Record Dates: First submitted 2020-10-27; First posted 2020-11-10 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
Keywords: Antibody Drug Conjugate; Phase 1/2; Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose Escalation - Schedule A: IMGC936 0.5 mg/kg (Experimental): Participants received IMGC936 0.5 milligrams (mg)/kilogram (kg) via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Escalation - Schedule A: IMGC936 1.0 mg/kg (Experimental): Participants received IMGC936 1.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Escalation - Schedule A: IMGC936 2.0 mg/kg (Experimental): Participants received IMGC936 2.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Escalation - Schedule A: IMGC936 4.0 mg/kg (Experimental): Participants received IMGC936 4.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Escalation - Schedule A: IMGC936 5.0 mg/kg (Experimental): Participants received IMGC936 5.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Escalation - Schedule A: IMGC936 6.0 mg/kg (Experimental): Participants received IMGC936 6.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Escalation - Schedule A: IMGC936 7.0 mg/kg (Experimental): Participants received IMGC936 7.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Escalation - Schedule B: IMGC936 2.0 mg/kg (Experimental): Participants received IMGC936 2.0 mg/kg on Days 1, 8, and 15 of a 28-day cycle for the first 2 cycles. On all subsequent cycles (Cycle 3 and beyond), participants received IMGC936 2.0 mg/kg on Days 1 and 8 of a 28-day cycle.
  Interventions: Drug: IMGC936
- Dose Expansion - NSCLC: IMGC936 6.0 mg/kg (Experimental): Participants received IMGC936 6.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936
- Dose Expansion - TNBC: IMGC936 6.0 mg/kg (Experimental): Participants received IMGC936 6.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
  Interventions: Drug: IMGC936

INTERVENTIONS:
Drug: IMGC936 — Antibody Drug Conjugate

SUMMARY:
This study is a Phase 1/2, first-in-human, open-label, dose-escalation, and expansion study designed to characterize the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary antitumor activity of IMGC936 administered by intravenous (IV) infusion.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation, and expansion study to determine the Maximum Tolerated Dose (MTD) and select the recommended Phase 2 dose (RP2D). Dose escalation follows a conventional 3+3 design; successive cohorts of 3 to 6 participants each will be evaluated in sequential escalating doses of single-agent IMGC936. Upon completion of the dose-escalation phase of the study, following determination of the RP2D, up to 5 expansion cohorts may be opened in tumor types selected from those enrolled in dose escalation.

Participants with relapsed or refractory, unresectable locally advanced or metastatic solid tumors including non-squamous non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC), colorectal cancer (CRC), gastroesophageal cancer, or pancreatic cancer will be enrolled.

IMGC936 is administered via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter, at the assigned dose for each cohort during dose escalation, and at the RP2D for expansion. Infusion duration will vary depending on dose and participant tolerability.

Sentinel dosing will be used for the first 2 dose levels of dose escalation. The first administration of IMGC936 in participants at the first 2 dose levels of dose escalation will be staggered by at least 48 hours. The dose-limiting toxicity (DLT) evaluation period is 21 days. Participants may continue on study drug until disease progression, adverse event (AE) requiring discontinuation, DLT during evaluation window, pregnancy, death, investigator decision, lost to follow up (LTFU), major protocol deviation requiring discontinuation, withdrawal of consent, or sponsor, investigator or regulatory agency terminates the study.

Tumor assessments are performed every 6 weeks (Q6W) while on study drug then every 12 weeks (Q12W). Tumor assessments continue until discontinuation criteria are met. If feasible, participants who discontinue study drug for reasons other than progressive disease (PD) (e.g., toxicity) should continue to undergo tumor assessments Q12W as post-treatment follow up until evidence of PD, initiation of another anticancer therapy, withdrawal of consent, LTFU, death, or end of study. Post-treatment follow up also includes following ongoing treatment emergent adverse events (TEAEs) until the event has resolved to baseline grade, the event is assessed by the investigator as stable, initiations of another anticancer therapy, withdrawal of consent, LTFU, death, or it has been determined that study drug or participation is not the cause of the AE.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with histologically proven, relapsed or refractory, unresectable locally advanced or metastatic non-squamous NSCLC, TNBC, CRC, gastroesophageal cancer, or pancreatic cancer for whom no therapy with demonstrated clinical benefit is available.

   1. NSCLC: Participants must have been treated with 1 to 4 prior lines of systemic therapy with no more than 2 chemotherapy containing lines.
   2. TNBC: Participants must have been treated with 1 to 4 prior lines of systemic therapy for metastatic disease, excluding adjuvant therapies.
   3. CRC: Participants must have been treated with 1 to 3 prior lines of systemic therapy.
   4. Gastroesophageal cancer: Participants must have been treated with 1 to 3 prior lines of systemic therapy.
   5. Pancreatic cancer: Participants must have been treated with 1 to 3 prior lines of systemic therapy, with no more than 2 chemotherapy containing lines.
2. Either measurable or non-measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and documented by computed tomography (CT) and/or magnetic resonance imaging (MRI) obtained within 28 days of Cycle 1 Day 1 (C1D1).

   * Dose escalation: Participants may have non-measurable or measurable disease
   * Dose expansion: Participants must have measurable disease
3. Age ≥ 18 years old.
4. Archival formalin-fixed paraffin-embedded (FFPE) tissue must be available. Participants may undergo a fresh tumor biopsy using a low risk, medically routine procedure to obtain a specimen for testing if a tumor sample is not available.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. If ECOG performance status is an inappropriate performance measurement for participant enrollment (for example, chronically non-ambulatory), then Karnofsky performance status must be ≥ 70.
6. Life expectancy ≥ 12 weeks.
7. Acceptable laboratory parameters as follows:

   * Platelet count ≥ 75 × 1000/microliter (μL) without transfusion within 28 days prior to initiation of study drug.
   * Absolute neutrophil count ≥ 1.5 × 1000/μL in the absence of any growth factor support within 21days prior to initiation of study drug.
   * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 3.0 × upper limit of normal (ULN); for participants with hepatic metastases, ALT and AST ≤ 5 × ULN.
   * Total bilirubin ≤ 1.5 × ULN, except participants with Gilbert's syndrome, who may enroll if the conjugated bilirubin is within normal limits.
   * Estimated glomerular filtration rate (eGFR) >30 milliliters (mL)/ minute (min)/1.73 square meter (m^2) or an estimated creatinine clearance of >30 mL/min.
   * Urinalysis protein and white occult blood cells within normal limits.
   * Negative serum pregnancy test for females of childbearing potential (FOCBP).
8. FOCBP, defined as not surgically sterilized (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) and between menarche and 1-year post menopause, must have a negative serum pregnancy test performed within 72 hours prior to initiation of study drug administration. Female participants must abstain from egg donation during the study.
9. FOCBP and male participants with partners of FOCBP must agree to use highly effective methods of contraception, from the time of consent through 28 weeks after discontinuation of study drug administration. Male participants must abstain from sperm donation during the study.
10. FOCBP is not pregnant or breastfeeding, or a male participant is not expecting to father children within the projected duration of the study, starting with screening visit through 28 weeks after the last dose of study drug.

Exclusion Criteria:

1. Active central nervous system (CNS) disease within the last 6 months.
2. Active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and/or monocular vision.
3. Participants who had prior therapies within the specified times below:

   * Systemic antineoplastic therapy at least 5 half-lives or 4 weeks (whichever is shorter) prior to initiation of study drug.
   * Mediastinal or pelvic radiation therapy within 6 weeks prior to initiation of study drug administration. Palliative, limited field radiation for symptom control to soft tissues, or bone lesions within 2 weeks prior to initiation of study drug.
4. Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities (except alopecia).
5. Clinically significant cardiovascular disease including but not limited to:

   * Myocardial infarction or unstable angina within 6 months prior to initiation of study drug.
   * Stroke or transient ischemic attack within 6 months prior to initiation of study drug.
   * Current clinically significant cardiac arrhythmias, for example, atrial fibrillation that are not well controlled with optimal medical intervention.
   * Current uncontrolled hypertension: systolic blood pressure > 160 millimeters of mercury (mmHg), diastolic blood pressure > 100 mmHg.
   * Current congestive heart failure (New York Heart Association class III-IV).
   * Current pericarditis or clinically significant pericardial effusion.
   * Current myocarditis.
   * Left ventricular ejection fraction (LVEF) of < 50% by scan
   * QTc interval > 480 milliseconds (msec)
6. Clinically significant pulmonary compromise, including pneumonia, pneumonitis, or a requirement for supplemental oxygen (excluding for sleep apnea) or history of ≥ Grade 3 drug-induced or radiation pneumonitis.
7. Serious concurrent illness or clinically relevant active infection, including, but not limited to the following:

   * Active hepatitis B or C infection (whether or not on active antiviral therapy).
   * Human immunodeficiency virus infection.
   * Cytomegalovirus infection.
   * Active COVID-19/SARS-CoV-2 infection. While SARS-CoV-2 testing is not mandatory for study entry, testing should follow local clinical practice guidelines/standards.
   * Any other concurrent infectious disease requiring IV antibiotics within 2 weeks prior to initiation of study drug.
8. History of prior bone marrow, stem cell, or solid organ transplantation.
9. Second primary invasive malignancy that has not been in remission for greater than 2 years except nonmelanoma skin cancer; cervical carcinoma in situ on biopsy; or squamous intraepithelial lesion on Pap smear; localized prostate cancer (Gleason score < 6); or resected melanoma in situ.
10. Major trauma or major surgery within 4 weeks prior to initiation of study drug.
11. Any serious underlying medical or psychiatric condition that would impair the ability of the participant to receive or tolerate the planned treatment at the study site.
12. Known hypersensitivity to any ingredient or any excipient contained in the drug formulation
13. Vaccination with any live virus vaccine within 4 weeks prior to initiation of study drug. Inactivated annual influenza vaccination is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CMO ImmunoGen, Study Director — ImmunoGen, Inc.
Locations (13):
- United States (7):
  - UCSD, La Jolla, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas
- Italy (3):
  - Policlinico di Modena, Modena
  - IRCCS Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Senese, Siena
- Spain (3):
  - START Madrid-FJD Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - START Madrid-HM CIOCC, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid

REFERENCES:
- [Derived] Scribner JA, Hicks SW, Sinkevicius KW, Yoder NC, Diedrich G, Brown JG, Lucas J, Fuller ME, Son T, Dastur A, Hooley J, Espelin C, Themeles M, Chen FZ, Li Y, Chiechi M, Lee J, Barat B, Widjaja L, Gorlatov S, Tamura J, Ciccarone V, Ab O, McEachem KA, Koenig S, Westin EH, Moore PA, Chittenden T, Gregory RJ, Bonvini E, Loo D. Preclinical Evaluation of IMGC936, a Next-Generation Maytansinoid-based Antibody-drug Conjugate Targeting ADAM9-expressing Tumors. Mol Cancer Ther. 2022 Jul 5;21(7):1047-1059. doi: 10.1158/1535-7163.MCT-21-0915. PMID 35511740

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a Dose Escalation and a Dose Expansion Phase.
Groups:
- Dose Escalation - Schedule A: IMGC936 0.5 mg/kg: Participants received IMGC936 0.5 milligrams (mg)/kilogram (kg) via intravenous (IV) infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
- Dose Escalation - Schedule B: IMGC936 2.0 mg/kg: Participants received IMGC936 2.0 mg/kg on Days 1, 8, and 15 of a 28-day cycle for the first 2 cycles. On all subsequent cycles (Cycle 3 and beyond), participants received IMGC936 3.0 mg/kg on Days 1 and 8 of a 28-day cycle.
- Dose Expansion - Non-small Cell Lung Cancer (NSCLC): IMGC936 6.0 mg/kg; Dose Expansion - Triple-negative Breast Cancer (TNBC): IMGC936 6.0 mg/kg: Participants received IMGC936 6.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
Period: Overall Study
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg | Dose Expansion - Non-small Cell Lung Cancer (NSCLC): IMGC936 6.0 mg/kg | Dose Expansion - Triple-negative Breast Cancer (TNBC): IMGC936 6.0 mg/kg
Started | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3 | 13 | 6
Received at Least 1 Dose of Study Drug | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3 | 13 | 6
Completed (Participants were considered "Completed" when discontinuation criteria were met.) | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3 | 13 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- Dose Escalation - Schedule A: IMGC936 0.5 mg/kg: Participants received IMGC936 0.5 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg | Dose Expansion - TNBC: IMGC936 6.0 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3 | 13 | 6 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (5.51) | 53.3 (8.39) | 59.3 (4.93) | 67.7 (5.69) | 61.3 (9.81) | 60.4 (7.63) | 63.4 (8.46) | 61.0 (5.57) | 64.8 (8.80) | 55.8 (10.96) | 61.1 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 2 | 6 | 6 | 32
  Male | 1 | 1 | 0 | 1 | 0 | 7 | 6 | 1 | 7 | 0 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  White | 3 | 2 | 2 | 2 | 3 | 9 | 9 | 3 | 11 | 5 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as any AEs with onset date between the first dose of IMGC936 and date of the last dose of IMGC936 + 30 days (inclusive) or date of the first anti-cancer therapy, whichever was earlier. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to approximately 3 years
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3
Participants
  Any TEAEs | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3
  SAEs | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 2

2. Primary Outcome: Dose Escalation Phase: Number of Participants With Dose-limiting Toxicities (DLTs) Based on National Cancer Institute (NCI) Common Terminology Criteria for AEs Version 5.0 (CTCAE v5.0)
Description: DLTs were defined based on TEAEs or abnormal laboratory values that met DLT criteria. Hematologic DLT: Grade 4 neutropenia lasting >7 days; ≥Grade 3 febrile neutropenia Grade 4 thrombocytopenia; Grade 3 thrombocytopenia associated with bleeding; ≥Grade 3 hemolysis. Non-hematologic DLT: Any ≥Grade 3 non-hematologic event, including Grade 3 ocular symptoms and signs; Grade 2 AEs that were prolonged inordinately; • Hepatic laboratory abnormalities meeting Hy's law criteria; Eye pain or reduction in visual acuity that did not respond to topical ophthalmic therapy. Hepatic DLT: Any elevation of ≥1 transaminases >8 * upper limit of normal (ULN); Any Grade 3 elevation of ≥1 transaminases >5.0-8.0 * ULN that did not resolve to Grade 2 within 7 days and Grade 1 within 14 days; Grade 3 elevation of total bilirubin >5 * ULN; Any Grade 3 elevation of total bilirubin >3.0-5.0 * ULN that did not resolve to Grade 2 within 7 days and Grade 1 within 14 days; Any event meeting criteria for Hy's law.
Time Frame: Cycle 1 (21 days for Schedule A and 28 days for Schedule B)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Dose Expansion Phase: Objective Response Rate (ORR) - Percentage of Participants With Objective Response as Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR: At least 30% decrease in the sum of the longest diameters (SoD) of target lesions, taking as reference the baseline SoD.
Time Frame: Up to approximately 3 years
Population: Response evaluable population included all participants who received at least 1 dose of study drug, had baseline measurable or non-measurable disease, and had at least 1 post-baseline radiographic tumor assessment or discontinued study drug due to clinical progression or death if no post-baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg | Dose Expansion - TNBC: IMGC936 6.0 mg/kg
Number analyzed (Participants) | 13 | 6
percentage of participants | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Dose Escalation and Dose Expansion Phase: Maximum Study Drug Concentration (Cmax)
Time Frame: Schedule A: Cycle 1 Day 1 (C1D1), C3D1; Schedule B: C1D1, C1D15
Population: The Pharmacokinetics Analysis Set (PAS) included all participants who received at least one dose of IMGC936 and from whom results of plasma or serum concentrations were obtained for at least one sampling point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (μg/mL)
Groups:
- Dose Escalation - Schedule A and Dose Expansion: IMGC936 6.0 mg/kg: Participants received IMGC936 6.0 mg/kg via IV infusion on Day 1 of Cycle 1 and every subsequent 21-day cycle thereafter.
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A and Dose Expansion: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 29 | 9 | 3
micrograms/milliliter (μg/mL)
  C1D1 | 14.17 (22) | 22.21 (5.6) | 56.69 (14.2) | 107.2 (9.6) | 114.8 (30.7) | 149.5 (21.6) | 162.4 (23.7) | 51.74 (9.8)
  C1D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  C1D15 |  |  |  |  |  |  |  | NA (NA) — Not calculable due to insufficient number of valid PK parameters
  C3D1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 8 | 1 | 0
  C3D1 | NA (NA) — Not calculable due to insufficient number of valid PK parameters |  | NA (NA) — Not calculable due to insufficient number of valid PK parameters |  | NA (NA) — Not calculable due to insufficient number of valid PK parameters | 168.4 (16.4) | NA (NA) — Not calculable due to insufficient number of valid PK parameters |

5. Secondary Outcome: Dose Escalation and Dose Expansion Phase: Number of Participants With Antidrug Antibodies (ADA)
Time Frame: Up to approximately 3 years
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg | Dose Expansion - TNBC: IMGC936 6.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3 | 13 | 6
Participants | 3 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 1

6. Secondary Outcome: Dose Escalation Phase: ORR - Percentage of Participants With Objective Response as Assessed by the Investigator Using RECIST v1.1
Description: ORR was defined as percentage of participants with a confirmed BOR of CR or PR. CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least 30% decrease in the SoD of target lesions, taking as reference the baseline SoD.
Time Frame: Up to approximately 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Dose Escalation and Dose Expansion Phase: Duration of Response (DOR) as Assessed by the Investigator Using RECIST v1.1
Description: DOR was defined as the time from the date of the first response (CR or PR), until the date of progressive disease (PD) or death from any cause, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase. DOR was estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 3 years
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg | Dose Expansion - TNBC: IMGC936 6.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 9 | 3 | 13 | 6
months | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated. | NA [NA to NA] — No participant had response; hence, data could not be calculated.

8. Secondary Outcome: Dose Expansion Phase: Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1
Description: PFS was defined as the time from initiation of study drug until the date of PD or death whichever occurred first, estimated using the Kaplan-Meier method. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to approximately 3 years
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg | Dose Expansion - TNBC: IMGC936 6.0 mg/kg
Number analyzed (Participants) | 13 | 6
months | 2.7 [0.7 to 6.7] | 1.2 [0.0 to 2.4]

9. Secondary Outcome: Dose Expansion Phase: Number of Participants With TEAEs, SAEs, and IMGC936 Related TEAEs That Led to Discontinuation
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as any AEs with onset date between the first dose of IMGC936 and date of the last dose of IMGC936 + 30 days (inclusive) or date of the first anti-cancer therapy, whichever was earlier. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to approximately 3 years
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg | Dose Expansion - TNBC: IMGC936 6.0 mg/kg
Number analyzed (Participants) | 13 | 6
Participants
  Any TEAEs | 13 | 6
  SAEs | 4 | 2
  IMGC936 related TEAEs That Led to Discontinuation | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Description: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg | Dose Expansion - TNBC: IMGC936 6.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 0/3 | 1/3 | 1/10 | 2/9 | 1/3 | 3/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 0/3 | 1/3 | 1/10 | 4/9 | 2/3 | 4/13 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 10/10 | 9/9 | 3/3 | 13/13 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg (N=10) | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg (N=9) | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg (N=3) | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg (N=13) | Dose Expansion - TNBC: IMGC936 6.0 mg/kg (N=6)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mycotic endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation - Schedule A: IMGC936 0.5 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 1.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 2.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 4.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 5.0 mg/kg (N=3) | Dose Escalation - Schedule A: IMGC936 6.0 mg/kg (N=10) | Dose Escalation - Schedule A: IMGC936 7.0 mg/kg (N=9) | Dose Escalation - Schedule B: IMGC936 2.0 mg/kg (N=3) | Dose Expansion - NSCLC: IMGC936 6.0 mg/kg (N=13) | Dose Expansion - TNBC: IMGC936 6.0 mg/kg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 5 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Cornea verticillata (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corneal epithelial microcysts (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 5 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 4 | 1 | 2 | 2
Keratopathy (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 2 | 2 | 6 | 7 | 2 | 8 | 4
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 3 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 4 | 1 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Sensation of blood flow (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Embolism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular disorders (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 1 | 0
Amylase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT04622774/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT04622774/SAP_001.pdf